CLINICAL TRIAL: NCT04349956
Title: Long-Term Follow-Up Study of Patients With Moderate to Severe, Painful Osteoarthritis of the Knee Who Participated in a Randomized, Placebo-Controlled Study of UBX0101
Brief Title: Long-Term Follow-Up Study of Patients With Osteoarthritis of the Knee Treated With UBX0101 or Placebo
Status: Terminated | Type: Observational
Why Stopped: Inability to achieve primary or secondary study objectives
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: UBX0101-05
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Painful Osteoarthritis; Osteoarthritis, Knee; Senescence
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients from a randomized placebo-controlled study of UBX0101: Patients with moderate to severe, painful OA of the knee who participated in a randomized, placebo-controlled study of UBX0101.
  Interventions: Drug: UBX0101 or placebo

INTERVENTIONS:
Drug: UBX0101 or placebo — This is an observational study. No intervention is administered.

SUMMARY:
A follow-up study to assess the long-term safety of intra-articular (IA) administration of UBX0101 in patients with painful knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This is a blinded, multi-center study to provide approximately 1 additional year of follow-up for patients with knee OA who participated in a randomized placebo-controlled study of IA UBX0101. No intervention is planned and patients will have 4 scheduled visits to collect follow-up assessments. The primary objective is to evaluate long-term safety and tolerability of IA administration of UBX0101 in patients with painful knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee OA who have completed a randomized placebo-controlled study of UBX0101.
* Patients who are willing and able to consent to having blinded, long-term follow-up; consent via legally authorized representative is not accepted.

Exclusion Criteria:

* Patients with any condition that, in the opinion of the Investigator, would likely interfere with adhering to the study schedule of visits for 12 months.
* Patients who are scheduled to undergo knee arthroplasty on either knee during the study.
* Patients who anticipate arthroscopic surgery on either knee at any time during the study.
* Patients who plan to receive treatment with an anti-nerve growth factor agent during the study.
* Patients who plan to participate in another investigational study (including interventional studies of investigational drugs and investigational treatments [e.g., braces, stem cells, and procedures]) during the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe painful knee OA who participated in a randomized, placebo-controlled study of UBX0101 and who consent to having blinded follow-up at the study site for 1 additional year of follow-up. Patients are permitted to take standard-of-care, background medications for OA.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events up to 1 additional year of follow up. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — UNITY Biotechnology
Locations (17):
- United States (17):
  - Coastal Clinical Research, LLC., Mobile, Alabama
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Biosolutions Clinical Research Center, La Mesa, California
  - Diablo Clinical Research, Walnut Creek, California
  - Well-Pharma Medical Research, Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Premier Medical Associates, The Villages, Florida
  - Chicago Clinical Research Institute, Chicago, Illinois
  - The Alliance for Multispecialty Research, Wichita, Kansas
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arcis Healthcare LLC dba Lowcountry Orthopaedics and Sports Medicine, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No